CLINICAL TRIAL: NCT06597240
Title: At-home Monitoring of Patients During Chemoradiation for Oesophageal CanceR: the AMCOR Trial
Brief Title: Home Monitoring During Chemoradiation
Acronym: AMCOR
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry); Nova Biomedical (Industry)
Responsible Party: Sponsor
Other Study IDs: PaNaMa nr. 11386
Record Dates: First submitted 2023-01-17; First posted 2024-09-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Oesophageal Cancer
Keywords: at-home monitoring; chemoradiation; oesophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AMCOR: Patients >18 years with locally advanced oesophageal cancer requiring chemoradiotherapy with curative intent.
  Interventions: Device: AMCOR

INTERVENTIONS:
Device: AMCOR — Participants will collect biometric and quality of life data for 9 or 10 weeks at home, depending on treatment schedule. Continuous step counting will be used to register physical activity. Participants will be asked to measure their blood pressure, heart rate, oxygen saturation level, pain level and temperature each morning, and weight 3 times a week. These measurements consume little time and are not harmful. Once a week they will perform a finger stick test themselves to determine creatinine concentration in the blood. In addition, patients fill in three questionnaires at four time points which will take approximately 20 minutes to complete per time point. We do not foresee reasonable risks of these diagnostic procedures for the participants.

SUMMARY:
Chemoradiotherapy is part of standard treatment for patients with locally advanced oesophageal cancer. Some patients with oesophageal cancer treated with chemoradiotherapy do not complete treatment due to toxicity, or face complications after treatment. Therefore, there is a need for better tools for assessing patients' fitness for chemoradiotherapy and to pick up early signals of deteriorating overall physical condition and complications during and after treatment to timely implement supportive care measures. Tools enabling monitoring physical activity, vital parameters and creatinine concentration in the blood at home are available but have not yet been implemented in patients undergoing chemoradiotherapy for oesophageal cancer. The feasibility and added value remain unknown.

DETAILED DESCRIPTION:
This is an observational feasibility study in which 30 ambulant patients with oesophageal cancer are continuously monitored from 1 week before chemoradiation until 3 weeks after chemoradiation for oesophageal cancer in addition to standard care.

We provide them with a monitoring kit of Siemens and a finger prick test of Nova Biomedical.

The monitoring kit of Siemens Healthineers contains multiple measuring tools, including:

* a blood pressure measuring device, which will be applied to the upper arm.
* an oxygen saturation measuring device, which will also measure the pulse when applied to the fingertip.
* a scale which will measure body weight.
* a skin thermometer which will detect body temperature.
* An activity tracker/watch which will measure every step taken during the day when worn around the wrist by the participant. All measurements will be automatically send to the online portal, which can be seen by the investigators.

Participants will receive a dedicated smartphone with an application to monitor their measurements at home for the duration of their study participation. The telephone does not provide any other functions than the specific app function.

With a finger stick test participants will measure the creatinine level in the blood. Nova Max Pro™ Creat Meter is a handheld analyser and miniaturized, single-use biosensor for whole blood creatinine testing. It enables assessment of renal function by fingerstick capillary blood sampling at home. It uses 1.2 μL capillary blood and shows the result in 30 seconds on the screen in μmol/L. The patient will carry out this measurement once a week the day before routine blood testing in the hospital. The values are transferred to the app via a Bluetooth® connection.

We will collect information on quality of life (QoL) and taste before, during and after treatment using a Quality of Life Questionnaire (QLQ) and a taste questionnaire. For QoL we will use the validated questionnaires of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, the core instrument that consists of 30 questions and the QLQ-OES18, the oesophageal cancer module that consists of 18 questions. The QLQ-OES18 consists of four scales, i.e., dysphagia, eating, reflux and pain and six single items, being swallowing saliva, choking when swallowing, dry mouth, taste problems, coughing and speech problems. The QLQ-C30 questionnaire consists 30 items and questions the overall global health status/QoL score, with the use of five functioning scores (physical, role, emotional, cognitive, and social functioning) and three composite symptom scores (fatigue, nausea, and vomiting). Six single-symptom items are also assessed being pain, dyspnea, insomnia, appetite loss, constipation, and diarrhea. The overall global health status and overall QoL score uses a seven-point Likert scale ranging from 'very poor' to 'excellent', and the remaining items in the EORTC use a four-point Likert scale ranging from 'not at all' to 'very much'. These scale scores are linearly converted to a 0-100 scale, where higher scores of the functioning scores and global QoL reflect higher levels of functioning and for the symptom scales higher scores reflect higher levels of symptom burden. Patients who reported 'a little' change for better or worse on a particular scale (function or symptom) had QLQ-C30 changes about 5 to 10. Those reporting 'moderate' change had changed about 10 to 20, and 'very much' change corresponded to a change greater than 20. A difference of 10 points up or down is often chosen as a clinically significant difference.

Taste will be assessed with the 'Chemotherapy-induced Taste Alteration Scale (CiTAS)'. This validated questionnaire consists of 18 questions with a Likert scale '1' to '5' (where '1' = no difficulty or absence of the disturbance and '5' = maximum difficulty or disturbance). It was developed based on semi-structured interviews with eight patients with cancer undergoing chemotherapy and is the first validated questionnaire regarding taste changes, available in many languages. It evaluates four dimensions of taste alterations: intensity of taste, discomfort, phantogeusie and parageusia, and general alterations of taste. The final score can be calculated by dividing the total score by the number of questions per section or in total, which gives an aim of the severity of the taste changes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at the time of signing informed consent.
* Histologically proven adenocarcinoma, squamous cell carcinoma or mixed type of the oesophagus or gastro-oesophageal junction.
* Indication for definitive or neoadjuvant CRT, with chemotherapy that consists of weekly carboplatin/paclitaxel.
* Written, informed consent.
* Ability to comply with all protocol required actions (at home measurements are done individually by the participant him- or herself).

Exclusion Criteria:

- Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent or the carrying out of the measurements at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck carcinoma eligible for chemoradiation with a curative intent, and chemotherapy that consists of cisplatin will be included in this study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of at home monitoring in addition to standard of care | From one week before the start of treatment until three weeks after the end of treatment
  To determine the feasibility of at home monitoring in addition to standard care of patients with oesophageal cancer during chemoradiotherapy. Feasible is defined as ≥80% of measurements completed in ≥80% of the patients.

SECONDARY OUTCOMES:
Determine completion rates | From one week before the start of treatment until three weeks after the end of treatment
  Determine completion rates per type of measurement
Determine the number of extra hospital visits | From one week before the start of treatment until three weeks after the end of treatment
  Determine the number of extra hospital visits triggered by home measurements.
Determine the number of extra telephone contacts | From one week before the start of treatment until three weeks after the end of treatment
  Determine the number of extra telephone contacts triggered by home measurements, subdivided by patient-initiated and nurse-initiated calls
Determine radiotherapy and chemotherapy completion rates | From one week before the start of treatment until three weeks after the end of treatment
  Determine radiotherapy and chemotherapy completion rates
Assess changes in quality of life from baseline in the domains overall health/QoL score, dysphagia and fatigue of the validated EORTC QLQ-C30 and QLQ-OES18. | From one week before the start of treatment until three weeks after the end of treatment
  The QLQ-OES18 consists of four scales, i.e., dysphagia, eating, reflux and pain and six single items, being swallowing saliva, choking when swallowing, dry mouth, taste problems, coughing and speech problems. The QLQ-C30 consists 30 items and questions the global health status/QoL, with the use of five functioning scores (physical, role, emotional, cognitive, and social functioning) and three symptom scores (fatigue, nausea, and vomiting). Six single-symptom items are also assessed being pain, dyspnea, insomnia, appetite loss, constipation, and diarrhea. The global health status and QoL score uses a seven-point Likert scale ranging from 'very poor' to 'excellent', and the remaining items in the EORTC use a four-point Likert scale ranging from not at all to very much. These scores are linearly converted to a 0-100 scale, where higher scores of the functioning scores and global QoL reflect higher levels of functioning and for the symptom scores reflect higher levels of symptom burden.
Assess taste changes from baseline with the use of Chemotherapy-induced Taste Alteration Scale (CiTAS) questionnaire | From one week before the start of treatment until three weeks after the end of treatment
  Assess taste changes from baseline with the Chemotherapy-induced Taste Alteration Scale (CiTAS), which consists of 18 questions with a Likert scale of 1 to 5 (where 1 = no difficulty or absence of the disturbance and 5 = maximum difficulty or disturbance). The final score can be calculated by dividing the total score by the number of questions per section or in total, which gives an aim of the severity of the taste changes.
Assess changes in quality of life from baseline in the remaining symptoms and domains of the EORTC QLQ-C30 and the oesophageal cancer specific EORTC QLQ-OES18. | From one week before the start of treatment until three weeks after the end of treatment
  The QLQ-OES18 consists of four scales, i.e., dysphagia, eating, reflux and pain and six single items, being swallowing saliva, choking when swallowing, dry mouth, taste problems, coughing and speech problems. The QLQ-C30 consists 30 items and questions the global health status/QoL, with the use of five functioning scores (physical, role, emotional, cognitive, and social functioning) and three symptom scores (fatigue, nausea, and vomiting). Six single-symptom items are also assessed being pain, dyspnea, insomnia, appetite loss, constipation, and diarrhea. The global health status and QoL score uses a seven-point Likert scale ranging from 'very poor' to 'excellent', and the remaining items in the EORTC use a four-point Likert scale ranging from not at all to very much. These scores are linearly converted to a 0-100 scale, where higher scores of the functioning scores and global QoL reflect higher levels of functioning and for the symptom scores reflect higher levels of symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf S.N. Fehrmann, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands